CLINICAL TRIAL: NCT03126045
Title: SPPLAASH Study : a Randomized Study Aiming at Evaluating the Incidence of Post Lumbar Puncture Headache (PLPH) With the Use of Atraumatic Needles in Hematology
Brief Title: A Randomized Study Evaluating the Incidence of Post Lumbar Puncture Headache With Atraumatic Needles in Hematology
Acronym: SPPLAASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-0302; 2017-A00915-48 (Other: ANSM)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Leukemia; Lymphoma
Keywords: Lumbar puncture; Post lumbar puncture headache; Atraumatic needle; Haematology
MeSH Terms: conditions — Leukemia; Lymphoma; Post-Dural Puncture Headache

STUDY DESIGN:
Intervention Model Description: Arm 1: standard needle Arm 2: Atraumatic needle
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither patients know the needle used during the spinal punction, nor the person collecting the information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard needle (Active Comparator): Patients perform a spinal punction according to the usual practice, with a standard needle.
  Interventions: Device: Standard needle
- Atraumatic needle (Experimental): Patients perform a spinal punction according to the usual practice, with an atraumatic needle.
  Interventions: Device: Atraumatic needle

INTERVENTIONS:
Device: Standard needle — Patients will perform a spinal punction with a standard needle, used in the usual practice. The standard needles have the following characteristics : BD 22 G x 3 ½ in, 90mm, Quincke spinal needle, Black hub.
  When more than 2 attempts for lumbar puncture fail, the investigator will proceed with standard techniques (BD 20G x 3 ½ in, Quincke spinal needle, 90mm, yellow hub). This is a failed lumbar puncture.
  Other Names: BD Yale 405256
  Arms: Standard needle
Device: Atraumatic needle — Patients will perform a spinal punction with an atraumatic needle, used in the hematological service of the CHU of Saint-Etienne. The atraumatic needles have the following characteristics : Vygon 24 G × 3 ½ in, 90mm, Whitacre Pencil Point Spinal Needle, Purple hub.
  When more than 2 attempts for lumbar puncture fail, the investigator will proceed with standard techniques (BD 20G x 3 ½ in, Quincke spinal needle, 90mm, yellow hub). This is a failed lumbar puncture.
  Other Names: Vygon 181.95
  Arms: Atraumatic needle

SUMMARY:
Lumbar punctures are implemented for the diagnosis of patients with hematologic symptoms as well as for the intrathecal chemotherapy injections. Post lumbar puncture headache is a common complication for patients and is characterized by the occurrence of a headache with an orthostatic component, with additional symptoms such as nausea. Some studies in neurology, anesthesia and gynecology have previously shown a decreased incidence for post lumbar puncture headache while using atraumatic needles as compared to standard needles. In this context, it is necessary to better document the incidence of post lumbar puncture headache with the use of atraumatic needles in hematologic patients.

DETAILED DESCRIPTION:
Lumbar punctures (LP) are implemented for the diagnosis of patients with hematologic symptoms as well as for the intrathecal chemotherapy injections. Post lumbar puncture headache (PLPH) is a common complication in around 30% of patients. PLPH is characterized by the occurrence of a headache with an orthostatic component within 12-72 hours after LP with additional symptoms such as nausea. Even if this phenomenon spontaneously resolves within 3 to 5 days, symptoms can immobilize the patient and can interfere with his daily activities. Technical procedures largely influence the incidence of PLPH. Indeed, some studies in neurology, anesthesia and gynecology have previously shown a decreased incidence for PLHP while using atraumatic needles as compared to standard needles. So far, few data are available for hematology. In this context, it is necessary to better document the incidence of PLPH with the use of atraumatic needles in hematologic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic syndromes undergoing a diagnostic lumbar puncture
* Signed written informed consent form
* Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

* Any known contraindication for the lumbar puncture procedure: increased intracranial pressure, blood clotting disorder, thrombocytopenia
* Any known infection
* Patient with a Body Mass index < 18 or Body Mass index > 40
* Any patient that requires an ultrasound guided lumbar puncture
* Patient that underwent a lumbar puncture within 6 months
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent (art. L.1121-6, L.112-7, L.1211-8, L.1211-9)
* Refusing participation
* Pregnancy or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Number of headache | 5 days
  Incidence of patients with mild and severe headache within 5 days following lumbar puncture as evaluated by verbal rating scales (intensity score ≥4) will be reported.

SECONDARY OUTCOMES:
Intensity of headache | 5 days
  Maximum intensity of headache as evaluated by verbal rating scale (scoring from 0 to 10) within 5 days following lumbar puncture will be reported for each patient.
Duration of significant headache | 5 days
  Duration in days of mild and severe headache (verbal rating scale score ≥ 4) within 5 days following lumbar puncture will be reported for each patient.
Pain intensity | 5 days
  Local and immediate Intensity Pain during lumbar puncture will be reported for each patient. Intensity is evaluated by verbal rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Guyotat, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No